CLINICAL TRIAL: NCT03248011
Title: Comparative Effectiveness of Hamstring Muscle Strain Injury Prevention Programs
Brief Title: Hamstring Strain in High School Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: General Electric (Industry); TRIA Orthopaedic Center (Other)
Responsible Party: Principal Investigator, Nathan D. Schilaty, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-003905
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Strains Thigh
Keywords: hamstring; ultrasound; intervention
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, repeated measures single- blind clinical trial.
Who Masked: Investigator
Masking Description: Group assignment will be masked to investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flexibility (Experimental): Stretching exercise
  Interventions: Other: Stretching
- Strength (Experimental): Eccentric hamstring strengthening exercise
  Interventions: Other: Strengthening
- Neuromuscular (Experimental): Balance exercise
  Interventions: Other: Neuromuscular
- Control (No Intervention): No exercise

INTERVENTIONS:
Other: Stretching — Lower extremity flexibility exercises will be performed
  Arms: Flexibility
Other: Strengthening — Eccentric hamstring strengthening exercises will be performed
  Arms: Strength
Other: Neuromuscular — Dynamic lower extremity balance and movement control exercises will be performed
  Arms: Neuromuscular

SUMMARY:
The purpose of the current study is, 1) Determine the effectiveness of injury prevention programs for prevention of hamstring muscle strains, 2) Identify how these programs impact athletes' flexibility, muscle stiffness, strength, and power, and 3) Determine the ability of a state-of-the-art imaging technology, shear wave elastography to predict future hamstring muscle strain injury.

DETAILED DESCRIPTION:
Hamstring strains are a significant problem for basketball athletes across levels of play for both sexes. The impact of hamstring muscle strains (HSMS) is significant. Injuries typically result in persistent symptoms and lengthy recovery periods which limit the athlete's practice and play time. Even more significantly, HSMS have high rates of reinjury. It is estimated that approximately one-third of hamstring strains are recurrent. Given the high incidence of HSMS and the substantial tendency for injuries to recur, it has been advocated the greatest impact may be achieved by the development of improved techniques for prevention of initial injury.

Multiple risk factors for HSMS have been identified. Perhaps the strongest modifiable risk factor associated with HSMS is an imbalance between quadriceps and hamstring strength, specifically the eccentric hamstrings and concentric quadriceps strength ratio. The rationale is that sufficient eccentric capacity of the hamstring muscles is necessary to offset the concentric quadriceps contraction during the terminal swing phase of running. Not surprisingly, prevention programs that emphasize eccentric hamstring strengthening have been effective in reduction of HSMS injury rates.Prospective studies have demonstrated mixed results regarding the relationship between hamstring flexibility and hamstring injury, and the effectiveness of a flexibility program for reduction of the incidence of HSMS remains controversial. Stretching duration, frequency, timing of stretching relative to sports activities and the type of stretch being performed have been suggested as important factors in the effectiveness of a flexibility program at reducing injury occurrence. In addition, reduced hip flexor and quadriceps flexibility has been identified as a risk factor for HSMS. Further investigation is necessary to determine if a flexibility program that addresses both anterior and posterior thigh musculature reduces injury risk. The role of neuromuscular (NM) deficits as a risk factor in HSMS injuries is unclear. Inclusion of NM exercises in a six week training period improved lower extremity control and movement discrimination, which has been suggested to contribute to HSMS injury prevention. However, the impact of a NM injury prevention program on HSMS rates has not been established.

Sheer wave elastography (SWE) represents an emerging imaging technology. This real-time imaging technique evaluates the local mechanical properties of muscles. Thus, SWE has the potential to provide more sensitive insight into muscle stiffness than flexibility assessment. Recent studies have utilized this technique to evaluate the effect of lower extremity positioning on hamstring stiffness. The relationship between stiffness measures obtained using SWE and HSMS has not, however, been established.

Key gaps in knowledge regarding HSMS injury prevention programs remain. Most critically, the effectiveness of HSMS prevention programs among basketball athletes is unknown. Furthermore, the comparative effectiveness of eccentric, flexibility, and NM training for reduction of HSMS injuries is also unknown. Assessment of lower extremity strength, rate of power production, flexibility, and stiffness (captured with SWE) may elucidate the mechanisms underlying the effectiveness of injury prevention training, and aid in enhancement of injury prevention programs. Thus, the potential impact of this proposal is profound as our investigative team aims to fill these gaps in knowledge. Ultimately, the results of this study have the potential to 1) reduce injuries among basketball athletes and consequently enhance and lengthen athletic careers, 2) provide scientific rationale underlying the effects of HSMS injury prevention training, and 3) determine if a novel ultrasound imaging technique may be effective in determining risk for HSMS.

ELIGIBILITY:
Inclusion criteria:

* member of high school basketball team
* school agreement to participate in study

Exclusion criteria:

* inability to ambulate independently
* lower extremity or back surgery within 1 year of study enrollment
* presence of neurological disease

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects who sustain a hamstring strain | Duration of school basketball season, approximately 4 months
  Physician based diagnosis

SECONDARY OUTCOMES:
Change in thigh strength | Baseline and post school basketball season, approximately 4 months
  This will be measured using an isokinetic dynamometer
Change in hamstring stiffness | Baseline, post school basketball season, approximately 4 months
  This will be measured using sheer wave elastography
Change in lower extremity power | Baseline, post school basketball season, approximately 4 months
  This will be measured using force plates
Change in lower extremity hamstring flexibility | Baseline, post school basketball season, approximately 4 months
  Measured using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Schilaty, DC, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Subject identification (ID) and study data (test results, injuries) will be shared with study co-investigators at TRIA Orthopaedics
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Co-Investigators will have access to the data as it is collected, for the duration of the study.
Access Criteria: Secured file transfer protocols will be utilized to transfer files between investigators. Only study co-investigators may access study data.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials